CLINICAL TRIAL: NCT05469100
Title: A Phase 1, Open-Label, Parallel-Cohort, Single-Dose Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics of LOXO-292
Brief Title: A Study of Effect of Selpercatinib (LY3527723) in Participants With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17484; J2G-OX-JZJE (Other: Eli Lilly and Company); LOXO-RET-18023 (Other: Loxo Oncology, Inc.)
Record Dates: First submitted 2022-07-20; First posted 2022-07-21 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Healthy; Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Selpercatinib (Control; Normal Renal Function) (Experimental): Participants with normal renal function (estimated glomerular filtration rate greater than or equal to [eGFR ≥ 90 milliliters per minute (mL/min) per 1.73 square meters (m²)] received a single 160 milligrams (mg) oral dose of Selpercatinib on Day 1, administered in a fasted state.
  Interventions: Drug: Selpercatinib
- Selpercatinib (Mild Renal Impairment) (Experimental): Participants with mild renal impairment (eGFR between 60 and 90 mL/min/1.73 m²) received a single 160 mg oral dose of Selpercatinib on Day 1, administered in a fasted state.
  Interventions: Drug: Selpercatinib
- Selpercatinib (Moderate Renal Impairment) (Experimental): Participants with moderate renal impairment (eGFR between 30 and 60 mL/min/1.73 m²) received a single 160 mg oral dose of Selpercatinib on Day 1, administered in a fasted state.
  Interventions: Drug: Selpercatinib
- Selpercatinib (Severe Renal Impairment) (Experimental): Participants with severe renal impairment (eGFR less than (<) 30 mL/min/1.73 m² and not requiring hemodialysis) received a single 160 mg oral dose of Selpercatinib on Day 1, administered in a fasted state.
  Interventions: Drug: Selpercatinib

INTERVENTIONS:
Drug: Selpercatinib — Administered orally
  Other Names: LY3527723; LOXO-292

SUMMARY:
The main purpose of this study is to assess the amount of study drug that reaches the bloodstream and the time it takes for the body to get rid of it when given to participants with renal (kidney) impairment compared to healthy participants. The study will last up to 9 days, excluding screening.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Body mass index (BMI) ≥ 18.0 and ≤ 40.0 kilograms per meter squared (kg/m²) and had a minimum weight of at least 50 kg at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), and blood and urine laboratory test results that are acceptable for the study
* Female of non childbearing potential: must have undergone sterilization procedures at least 6 months prior to the Screening
* Males who are capable of fathering a child must agree to use contraception from the time of the dose administration through 6 months after the last dose

For renal participants:

* Participant has stable renal disease status and function at least 1 month prior to LOXO-292 administration.
* Participant is not currently or has not previously being on hemodialysis
* Baseline estimated glomerular filtration rate (eGFR) based on the Modification of Diet in Renal Disease (MDRD) equation at screening as follows:

  * Severe Renal Impairment (RI): < 30 milliliter per minute (mL/min)/1.73m²
  * Moderate RI: ≥ 30 and < 60 mL/min/1.73m²
  * Mild RI: ≥ 60 and < 90 mL/min/1.73m²

The MDRD equation is as follows (for females multiply result by 0.742, if African American multiply result by 1.212):

eGFR = 175 x [serum creatinine in milligrams per deciliter (mg/dL) measured with a standardized assay]^-1.154 x (Age)^-0.203

Exclusion Criteria:

For renal participants:

* Has rapidly fluctuating renal function, as determined by historical measurements; or has demonstrated or suspected renal artery stenosis. Rapidly fluctuating renal function is defined as creatinine clearance or eGFR that differs by more than 20% within at least 3 months of the screening creatinine clearance or eGFR. If historical measurements are not available, then the 2 screening measurements will be used to demonstrate stability.
* Participants who have had a renal transplant, a nephrectomy, or participants with a known history of nephrotic syndrome.
* Participants who have required new medication for renal disease within 30 days prior to Check-in

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - Anaheim Regional Center, Anaheim, California
  - Stanford Health Care, Valley Care Program, Pleasanton, California
  - Orange County Research Center, Tustin, California
  - Riverside Clinical Research, Edgewater, Florida
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Started | 13 | 9 | 8 | 7
Received at Least One Dose of Selpercatinib | 13 | 9 | 8 | 7
Completed | 13 | 9 | 8 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Selpercatinib (Control; Normal Renal Function): Participants with normal renal function (eGFR ≥ 90 mL/min/1.73 m²) received a single 160 mg oral dose of Selpercatinib on Day 1, administered in a fasted state.
- Selpercatinib (Severe Renal Impairment): Participants with severe renal impairment (eGFR < 30 mL/min/1.73 m² and not requiring hemodialysis) received a single 160 mg oral dose of Selpercatinib on Day 1, administered in a fasted state.
- Total: Total of all reporting groups
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment) | Total
Number analyzed (Participants) | 13 | 9 | 8 | 7 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.40 (6.42) | 58.40 (6.23) | 62.60 (6.02) | 61.30 (5.85) | 60.20 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 2 | 2 | 13
  Male | 7 | 6 | 6 | 5 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 1 | 3 | 11
  Not Hispanic or Latino | 9 | 6 | 7 | 4 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 3 | 4 | 2 | 16
  White | 6 | 6 | 4 | 5 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 9 | 8 | 7 | 37

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to the Last Observed Non-zero Concentration (AUC0-t) of Selpercatinib in Plasma
Description: PK: AUC0-t of Selpercatinib
Time Frame: Predose (within 30 minutes), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable PK data. Participants were excluded from the analysis if they experienced emesis (vomiting) that occurred at or before 2 times the median time to maximum observed plasma concentration (Tmax).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
nanogram*hour per milliliter (ng*hr/mL) | 19770 (52.1) | 23440 (36.0) | 29270 (25.6) | 20640 (71.0)

2. Primary Outcome: PK: Area Under the Concentration-time Curve, From Time 0 Extrapolated to Infinity (AUC0-inf) of Selpercatinib in Plasma
Description: PK: AUC0-inf of Selpercatinib
Time Frame: as for outcome 1
Population: All enrolled participants who received at least one dose of the study drug and had evaluable PK data. Participants were excluded from the analysis if they experienced emesis (vomiting) that occurred at or before 2 times the median Tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
nanogram*hour per milliliter (ng*hr/mL) | 19870 (52.0) | 23510 (36.0) | 29470 (25.8) | 21000 (71.4)

3. Primary Outcome: PK: Percentage of AUC0-inf Extrapolated (AUC%Extrap) of Selpercatinib.in Plasma
Description: PK: Percentage of AUC0-inf extrapolated was calculated as (1 - AUC0-t/AUC0-inf) * 100.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of AUCextrap
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
percentage of AUCextrap | 0.4856 (0.12819) | 0.2988 (0.10713) | 0.6738 (0.33398) | 1.706 (1.5917)

4. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of Selpercatinib in Plasma
Description: PK: Cmax of Selpercatinib
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
nanogram per milliliter (ng/mL) | 1399 (107.3) | 2247 (22.3) | 1742 (25.1) | 1006 (159.6)

5. Primary Outcome: PK: Time to Maximum Observed Plasma Concentration (Tmax) of Selpercatinib in Plasma
Description: PK: Tmax of Selpercatinib
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
hours (hr) | 1.500 [1.00 to 24.00] | 1.500 [1.50 to 2.00] | 1.500 [1.00 to 3.00] | 1.000 [0.50 to 24.00]

6. Primary Outcome: PK: Apparent First Order Terminal Elimination Rate Constant (Kel) of Selpercatinib in Plasma
Description: PK: Apparent terminal elimination rate constant; represents the fraction of drug eliminated per unit time calculated by linear least squares regression analysis using the maximum number of points in the terminal log linear phase (e.g., three or more non zero plasma concentrations).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: One per hour (1/hour)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
One per hour (1/hour) | 0.02853 (0.0043443) | 0.03434 (0.012429) | 0.02662 (0.0047866) | 0.02204 (0.0061504)

7. Primary Outcome: PK: Apparent First-order Terminal Elimination Half-life (t½) of Selpercatinib in Plasma
Description: PK: t½ of Selpercatinib.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
hours (hr) | 24.854 (4.0850) | 22.632 (8.7328) | 27.139 (7.1091) | 33.828 (10.4879)

8. Primary Outcome: PK: Apparent Total Plasma Clearance After Oral (Extravascular) Administration (CL/F) of Selpercatinib in Plasma
Description: PK: CL/F of Selpercatinib
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters per Hour (L/h)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
Liters per Hour (L/h) | 8.976 (4.6533) | 7.188 (2.6117) | 5.581 (1.3807) | 9.184 (6.5822)

9. Primary Outcome: PK: Apparent Volume of Distribution During the Terminal Elimination Phase After Oral (Extravascular) Administration (Vz/F) of Selpercatinib in Plasma
Description: PK: Vz/F of Selpercatinib
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
Liter | 334.5 (225.17) | 227.9 (106.14) | 219.4 (82.255) | 444.7 (309.92)

10. Primary Outcome: PK: Unbound AUC0-t (AUC0-t,u) of Selpercatinib in Plasma
Description: AUC0-t,u was calculated by multiplying AUC0-t by Fu (i.e., AUC0-t*Fu). Fu represented the unbound fraction of Selpercatinib in plasma, that is, the portion of the drug not bound to plasma proteins.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
nanogram*hour per milliliter (ng*hr/mL) | 533.1 (54.3) | 659.7 (24.4) | 856.3 (28.0) | 709.9 (93.0)

11. Primary Outcome: PK: Unbound AUC0-inf (AUC0-inf,u) of Selpercatinib in Plasma
Description: AUC0-inf,u was calculated by multiplying AUC0-inf by Fu (i.e., AUC0-inf*Fu). Fu represented the unbound fraction of Selpercatinib in plasma, that is, the portion of the drug not bound to plasma proteins.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
nanogram*hour per milliliter (ng*hr/mL) | 535.7 (54.3) | 661.6 (24.4) | 862.1 (28.1) | 722.3 (93.9)

12. Primary Outcome: PK: Unbound Cmax (Cmax,u) of Selpercatinib in Plasma
Description: Cmax,u was calculated by multiplying Cmax by Fu (i.e., Cmax*Fu). Fu represented the unbound fraction of Selpercatinib in plasma, that is, the portion of the drug not bound to plasma proteins.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
nanogram per milliliter (ng/mL) | 37.72 (113.6) | 63.23 (23.4) | 50.95 (28.5) | 34.60 (187.8)

13. Primary Outcome: PK: Unbound CL/F (CL/F,u) of Selpercatinib in Plasma
Description: CL/F,u was calculated by multiplying CL/F by Fu (i.e., CL/F*Fu). Fu represented the unbound fraction of Selpercatinib in plasma, that is, the portion of the drug not bound to plasma proteins.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters per Hour (L/h)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
Liters per Hour (L/h) | 337.9 (194.45) | 247.9 (58.030) | 191.6 (49.277) | 300.6 (294.31)

14. Primary Outcome: PK: Unbound Vz/F (Vz/F,u) of Selpercatinib in Plasma
Description: Vz/F,u was calculated by multiplying Vz/F by Fu (i.e., Vz/F*Fu). Fu represented the unbound fraction of Selpercatinib in plasma, that is, the portion of the drug not bound to plasma proteins.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter (L)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
Liter (L) | 12700 (9498.5) | 8214 (4487.5) | 7697 (3676.1) | 14340 (12842)

15. Primary Outcome: PK: Cumulative Amount of Selpercatinib Excreted (CumAe) in Urine
Description: PK: CumAe was reported. The urine sampling time points from pre-dose through 168 hours post-dose were used to assess this outcome.
Time Frame: Predose (spot collection), 4, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligram (mg)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
milligram (mg) | 16.14 (9.5297) | 14.54 (3.1611) | 13.94 (5.3203) | 7.652 (5.4210)

16. Primary Outcome: PK: Cumulative Percentage of Administered Selpercatinib Dose (Cum%Dose) Excreted in Urine
Description: PK: Cum%Dose was reported. The urine sampling time points from pre-dose through 168 hours post-dose were used to assess this outcome.
Time Frame: Predose (spot collection), 4, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of dose excreted
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
percentage of dose excreted | 10.09 (5.9560) | 9.087 (1.9757) | 8.713 (3.3252) | 4.782 (3.3881)

17. Primary Outcome: PK: Renal Clearance (CLr) of Selpercatinib in Urine
Description: PK: CLr of Selpercatinib was reported.The urine sampling time points from pre-dose through 168 hours post-dose were used to assess this outcome.
Time Frame: Predose (spot collection), 4, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliter per hour (mL/hr)
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
Number analyzed (Participants) | 10 | 8 | 8 | 7
milliliter per hour (mL/hr) | 735.9 (230.39) | 641.6 (243.96) | 480.4 (208.23) | 314.6 (94.084)

ADVERSE EVENTS:
Time Frame: Baseline up to 15 days
Description: All enrolled participants who received at least one dose of Selpercatinib.
Arm/Group | Selpercatinib (Control; Normal Renal Function) | Selpercatinib (Mild Renal Impairment) | Selpercatinib (Moderate Renal Impairment) | Selpercatinib (Severe Renal Impairment)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/9 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/9 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 2/13 | 3/9 | 3/8 | 3/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selpercatinib (Control; Normal Renal Function) (N=13) | Selpercatinib (Mild Renal Impairment) (N=9) | Selpercatinib (Moderate Renal Impairment) (N=8) | Selpercatinib (Severe Renal Impairment) (N=7)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT05469100/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT05469100/SAP_001.pdf